CLINICAL TRIAL: NCT02101788
Title: A Randomized Phase II/III Study to Assess the Efficacy of Trametinib (GSK 1120212) in Patients With Recurrent or Progressive Low-Grade Serous Ovarian Cancer or Peritoneal Cancer
Brief Title: Trametinib in Treating Patients With Recurrent or Progressive Low-Grade Ovarian Cancer or Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00629; NCI-2014-00629 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0281 (Other: NRG Oncology); GOG-0281 (Other: CTEP); P50CA083639 (NIH); U10CA180868 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Borderline Ovarian Serous Tumor; Micropapillary Serous Carcinoma; Ovarian Serous Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Ovarian Low Grade Serous Adenocarcinoma; Recurrent Primary Peritoneal Serous Adenocarcinoma
MeSH Terms: conditions — Cystadenocarcinoma, Serous | interventions — Letrozole; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Tamoxifen; Topotecan; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan) (Active Comparator): Patients receive clinician's choice of either letrozole PO QD on days 1-28, tamoxifen citrate PO BID on days 1-28, paclitaxel IV over 1 hour on days 1, 8, and 15, pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 1, or topotecan IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients developing progressive disease may cross over to Arm B.
  Interventions: Drug: Letrozole; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tamoxifen Citrate; Drug: Topotecan
- Arm B (trametinib) (Experimental): Patients receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Letrozole — Given PO
  Other Names: CGS 20267; CGS-20267; CGS20267; Femara; Fempro
  Arms: Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan)
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI 46474; ICI-46474; ICI46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide
  Arms: Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan)
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
  Arms: Arm A (letrozole, tamoxifen, paclitaxel, PLD, topotecan)
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras
  Arms: Arm B (trametinib)

SUMMARY:
This phase II/III trial studies how well trametinib works and compares it to standard treatment with either letrozole, tamoxifen, paclitaxel, pegylated liposomal doxorubicin, or topotecan in treating patients with low-grade ovarian cancer or peritoneal cavity cancer that has come back (recurrent), become worse (progressive), or spread to other parts of the body. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether trametinib is more effective than standard therapy in treating patients with ovarian or peritoneal cavity cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the progression-free survival (PFS) hazard ratio of trametinib compared to that of "commercially available therapies" consisting of one of five commercially available agents in women with recurrent low-grade serous carcinoma of the ovary or peritoneum previously treated with platinum-based chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the nature, frequency and maximum degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4 for each treatment arm.

II. To determine the quality of life, as assessed by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O).

IIa. To compare trametinib to the control arm with regard to patients' self-reported acute (up to post-cycle 6) quality of life as measured by the FACT-O-Trial Outcome Index (TOI).

IIb. To compare trametinib to the control arm with regard to patients' self-reported acute (up to post-cycle 6) neurotoxicity as measured by the FACT-Gynecologic Oncology Group (GOG)-Neurotoxicity (NTX).

III. To estimate the objective response rate (RR) of patients in each treatment arm.

IV. To test whether high expression of pERK, as quantified by immunohistochemistry (IHC), is associated with better prognosis (RR or PFS) among patients receiving the randomized treatment.

V. To test whether genetic changes associated with MAPK pathway activation (KRAS, NRAS, HRAS, BRAF, MEK, ERBB2 or NF1) are associated with improved prognosis (RR or PFS) among patients receiving the randomized treatment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive clinician's choice of either letrozole orally (PO) once daily (QD) on days 1-28, tamoxifen citrate PO twice daily (BID) on days 1-28, paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15, pegylated liposomal doxorubicin hydrochloride (PLD) IV over 1 hour on day 1, or topotecan IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients developing progressive disease may cross over to Arm B.

ARM B: Patients receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than 18 with the following tumors are included in the study:

  * Patients initially diagnosed with low-grade serous ovarian or peritoneal carcinoma that recur as low-grade serous carcinoma (invasive micropapillary serous carcinoma or invasive grade I serous carcinomas as defined by GOG, Federation of Obstetricians and Gynecologists [FIGO], World Health Organization [WHO] or Silverberg)
  * Patients initially diagnosed with serous borderline ovarian or peritoneal carcinoma that recur as low-grade serous carcinoma (invasive micropapillary serous carcinoma or invasive grade I serous carcinomas as defined by GOG, FIGO WHO or Silverberg)
* At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g. MAJOR: laparotomy, laparoscopy, thoracotomy, VATS [video assisted thorascopic surgery]); there is no restriction on MINOR procedures: (e.g. central venous catheter placement, ureteral stent placement or exchange, tumor core or fine-needle aspirate [FNA] biopsy)
* Patients must have documented low-grade serous carcinoma; confirmation must occur by prospective pathology review prior to study entry; the prospective pathology review can be done on tissue from the recurrent carcinoma or from original diagnostic specimen
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one target lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI; all imaging studies must be performed within 28 days prior to registration
* Prior therapy

  * Patients must have recurred or progressed following at least one platinum-based chemotherapy regimen
  * Patients may have received an unlimited number of prior therapy regimens
  * Patients may not have received all of the five choices in the "standard therapy" arm
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including chemotherapy and radiation therapy, must be discontinued at least 4 weeks prior to registration; any investigational agent must be discontinued at least 28 days prior to registration
* Trametinib, can cause fetal harm when administered to a pregnant woman; women of child-bearing potential (i.e. patients whose reproductive organs remain in place and who have not passed menopause) and men must agree to use a highly effective method of contraception (e.g. hormonal, intrauterine device or; abstinence*) prior to study entry, during the study participation, and for six months after the last dose of the drug; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to randomization, cannot be breast-feeding, and must agree to use a highly effective form of contraception throughout the treatment period and for 6 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * Abstinence is only acceptable when this is in line with the preferred and usual lifestyle of the patient
* Patients must have the ability to understand and sign an approved informed consent and authorization permitting release of personal health information
* Patients must have a GOG performance status of 0 or 1
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome, bowel obstruction, or major resection of the stomach or bowel
* All prior treatment-related toxicities must be CTCAE v4 grade =< 1 (except alopecia) at the time of randomization
* Patients must have a left ventricular ejection fraction >= lower limit of normal by echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min (within 14 days prior to treatment)
* Bilirubin =< 1.5 times upper limit of normal (within 14 days prior to treatment)
* Alanine aminotransferase (ALT) =< 2.5 times upper limit of normal (within 14 days prior to treatment)
* Aspartate aminotransferase (AST) =< 2.5 times upper limit of normal (within 14 days prior to treatment)
* Albumin >= 2.5 g/dL (within 14 days prior to treatment)
* Prothrombin time (PT) and activated partial thromboplastin time (APTT) =< 1.5 times upper limit of normal (within 14 days prior to treatment)
* Neutrophil count >= 1.5 x 10^9/L (within 14 days prior to treatment)
* Platelet count >= 100 x 10^9/L (within 14 days prior to treatment)
* Hemoglobin >= 9.0 g/dL (within 14 days prior to treatment)
* If letrozole is selected as the control therapy, patients must be postmenopausal, either following bilateral oophorectomy or at least 5 years after spontaneous menopause; patients within 5 years of spontaneous menopause or who have had a hysterectomy without bilateral oophorectomy must have postmenopausal luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels; patients on hormone replacement therapy (HRT) must agree to withdrawal of hormone therapy before letrozole is started

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib or standard of care agent
* If patients have had a potential index lesion radiated, it must have progressed post radiation therapy to be used as a measurable eligibility lesion
* Patients may not have received prior MEK, v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS), or v-raf murine sarcoma viral oncogene homolog B1 (BRAF) inhibitor therapy
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Patients may not be receiving any other anti-cancer or investigational agents
  * Because the composition, PK, and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* Patients with known leptomeningeal or brain metastases or spinal cord compression should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with a bowel obstruction or any other gastrointestinal condition that might affect absorption of the oral drug should be excluded; this would include patients with inability to swallow and retain orally-administered medication, malabsorption syndrome, or those with a major resection of the stomach or bowels
* Patients with a history of interstitial lung disease or pneumonitis
* Patients with a previous or current malignancy at other sites should be excluded, with the exception of:

  * Curatively treated local tumors such as carcinoma-in-situ of the cervix, basal or squamous cell carcinoma of the skin
  * Tumors for which no relapse has been observed within 5 years
* Known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients, or to dimethyl sulfoxide (DMSO), or to Cremophor EL (polyoxyethylated castor oil); please note, exclusion for Cremophor is unnecessary unless paclitaxel is the only agent available and the patient randomizes to the conventional therapy option
* Patients with a history or evidence of cardiovascular risk, including any of the following:

  * Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN)
  * Bazett's corrected QT (QTcB) >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias
  * Exception: Subjects with controlled atrial fibrillation for > 30 days prior to randomization are eligible
  * History of (within 6 months prior to randomization) acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting
  * History or evidence of current >= class II congestive heart failure as defined by New York Heart Association (NYHA)
  * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators or permanent pacemakers
  * Known cardiac metastases
* Patients with a history or current evidence/risk of retinal vein occlusion (RVO)
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Patients who require use of a concomitant medication that can prolong the QT interval
* Animal reproductive studies have not been conducted with trametinib; therefore, the study drug must not be administered to pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2025-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Gershenson, Principal Investigator — NRG Oncology
Locations (501):
- United States (488):
  - Tennessee Valley Gynecologic Oncology, Huntsville, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Sutter Davis Hospital, Davis, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Research Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- United Kingdom (13):
  - Bristol Royal Infirmary, Bristol, England
  - Addenbrookes Hospital-Medical School, Cambridge, England
  - Saint Bartholomew's Hospital, London, England
  - Hammersmith Hospital, London, England
  - University College London Hospital, London, England
  - Christie Hospital, Manchester, England
  - Musgrove Park Hospital, Somerset, England
  - Saint James's University Hospital, West Yorkshire, England
  - Belfast City Hospital, Belfast, Northern Ireland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Center, Glasgow, Scotland
  - The Royal Marsden NHS Foundation Trust-Chelsea, London
  - Nottingham City Hospital, Nottingham

REFERENCES:
- [Derived] Gershenson DM, Miller A, Brady WE, Paul J, Carty K, Rodgers W, Millan D, Coleman RL, Moore KN, Banerjee S, Connolly K, Secord AA, O'Malley DM, Dorigo O, Gaillard S, Gabra H, Slomovitz B, Hanjani P, Farley J, Churchman M, Ewing A, Hollis RL, Herrington CS, Huang HQ, Wenzel L, Gourley C. Trametinib versus standard of care in patients with recurrent low-grade serous ovarian cancer (GOG 281/LOGS): an international, randomised, open-label, multicentre, phase 2/3 trial. Lancet. 2022 Feb 5;399(10324):541-553. doi: 10.1016/S0140-6736(21)02175-9. PMID 35123694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 260 patients enrolled before accrual closed on 04/10/2018.
Groups:
- Arm A - Control Arm: Investigators choice of Letrozole 2.5 mg po qd continuously, tamoxifen 20mg po bid continuously, paclitaxel 80mg/m2 IV over 1 hr on day 1q 7d, 3 wks on, 1 wk off, Pegylated Liposomal Doxorubicin 40 or 50mg/m2 IV over 1 hr on day 1 q. 28d, Topotecan 4.0mg/m2 over 30 min on day 1,8 and 15 of a 28 day cycle. For each arm, 1 cycle - 28 days
- Arm B - Experimental Arm: Trametinib 2 mg po daily continuous treatment, For each arm, 1 cycle = 28 days
Period: Overall Study
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm
Started | 130 | 130
Crossover From Arm A to Arm B | 88 | 0
Completed | 120 | 116
Not Completed | 10 | 14

BASELINE CHARACTERISTICS:
Population: All enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.89 (14.03) | 53.57 (14.13) | 53.7 (14.1)
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 9 | 10 | 19
  30-39 years | 18 | 16 | 34
  40-49 years | 21 | 22 | 43
  50-59 years | 28 | 35 | 63
  60-69 years | 39 | 33 | 72
  >= 70 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 130 | 260
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 118 | 118 | 236
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 5 | 4 | 9
  White | 114 | 115 | 229
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 102 | 103 | 205
  United Kingdom | 28 | 27 | 55
Number of Prior Treatment Regimens [Count of Participants; unit: Participants]
  1 Prior Treatment Regimens | 30 | 29 | 59
  2 Prior Treatment Regimens | 37 | 39 | 76
  3 or More Prior Treatment Regimens | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) was defined as the number of months between study enrollment and documentation of disease progression (RECIST 1.1) or death from any cause. Patients still alive and disease free at the last followup were censored on the date of last CT Scan.Participants were analyzed based on their group of assignment. Patients on Arm A who progressed were permitted to receive Arm B treatment. Study time for Arm A patients who crossed over was not included in the PFS endpoint definition.
Time Frame: Time from study entry to time of progression or death, an average of 7 months for arm A and 13 months for arm B
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm
Number analyzed (Participants) | 130 | 130
months | 7.2 [5.6 to 9.9] | 13.0 [9.9 to 15.0]

2. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Number of treated patients with Adverse Events (grade 3 or higher) observed while receiving randomized therapy. Excludes AEs observed among control patients treated with trametinib after crossover.Participants were analyzed based on their group of assignment. Patients on Arm A who progressed were permitted to receive Arm B treatment. Study time for Arm A patients who crossed over was not included in the AE endpoint definition.
Time Frame: During treatment period and up to 100 days after stopping the study treatment
Population: Treated with randomized therapy
Measure: Number; unit: participants
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm
Number analyzed (Participants) | 127 | 127
participants
  Abdominal pain | 22 | 7
  Anemia | 12 | 16
  Diarrhea | 4 | 13
  Fatigue | 5 | 10
  Hypertension | 6 | 15
  Nausea | 14 | 12
  Neutrophil count decreased | 1 | 8
  Rash maculo-papular | 0 | 9
  Small Intestinal Obstruction | 9 | 16
  Vomiting | 10 | 9

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the number of months between study enrollment and death from any cause. Patients still alive at the last follow-up were censored on the date of last contact. Patients with disease progression on the Control arm were allowed to cross over to the trametinib arm. Per the protocol, the intent-to-treat OS analysis was not adjusted for crossover.
Time Frame: Time from study entry to time of death or date of last contact, an average of 29 months for arm A and 37 months for arm B
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm
Number analyzed (Participants) | 130 | 130
Months | 29.2 [23.5 to 51.6] | 37.0 [30.3 to NA] — insufficient number of participants with events

4. Secondary Outcome: Objective Tumor Response Rate (Complete Response and Partial Response)
Description: The Response Rates were estimated as the binomial proportion of patients with Best Overall Response of Complete or Partial response according to RECIST 1.1 criteria.
Time Frame: Time from study entry to time of progression or death, an average of 7 months for arm A and 13 months for arm B
Population: Randomized patients
Measure: Number; unit: participants
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm
Number analyzed (Participants) | 130 | 130
participants | 8 | 34

5. Secondary Outcome: Patients Reported Acute Quality of Life
Description: Patient reported quality of life was measured with the Treatment Outcome Index (TOI) of the Functional Assessment of Cancer Therapy for ovarian cancer (FACT-O TOI). The FACT-O TOI is a scale for assessing general QOL of ovarian cancer patients. It consists of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Ovarian Cancer subscale (11 items). . The FACT-O TOI score is calculated as the sum of the subscale scores if more than 80% of the FACT-O TOI items provide valid answers and all of the component subscales have valid scores. The FACT-O TOI score ranges 0-100 with a large score suggesting better QOL. Participants were analyzed based on their group of assignment. Patients on Arm A who progressed were permitted to receive Arm B treatment. Study time for Arm A patients who crossed over was not included in the quality of life endpoint definition
Time Frame: 1. baseline (prior to cycle 1), 12 weeks (prior to cycle 4), 24 weeks (4 weeks post cycle 6), 36 weeks post cycle 1, 52 weeks post cycle 1.
Population: Patients who provided baseline and ≥ 1 follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm A (Letrozole, Tamoxifen, Paclitaxel, PLD, Topotecan): Patients receive clinician's choice of either letrozole PO QD on days 1-28, tamoxifen citrate PO BID on days 1-28, paclitaxel IV over 1 hour on days 1, 8, and 15, pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 1, or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients developing progressive disease may cross over to Arm B.
  Letrozole: Given PO
  Paclitaxel: Given IV
  Pegylated Liposomal Doxorubicin Hydrochloride: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Tamoxifen: Given PO
  Tamoxifen Citrate: Given PO
  Topotecan: Given IV
  Topotecan Hydrochloride: Given IV
- Arm B (Trametinib): Patients receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Quality-of-Life Assessment: Ancillary studies
  Trametinib: Given PO
  Trametinib Dimethyl Sulfoxide: Given PO
Arm/Group | Arm A (Letrozole, Tamoxifen, Paclitaxel, PLD, Topotecan) | Arm B (Trametinib)
Number analyzed (Participants) | 98 | 100
score on a scale
  Baseline | 74.5 (16.6) | 74.5 (13.7)
  12 Weeks | 74.2 (16.0) | 70.6 (13.5)
  24 Weeks | 70.2 (15.5) | 73.0 (12.8)
  36 Weeks | 69.3 (18.6) | 72.6 (12.8)
  52 Weeks | 72.1 (16.9) | 73.3 (14.3)

6. Secondary Outcome: Patient Reported Acute Peripheral Neuropathy Symptoms
Description: Patient reported peripheral neuropathy symptoms was measured with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The FACT/GOG-Ntx subscale contains 4 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). According to the FACIT measurement system, the Ntx score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The Ntx score ranges 0-16 with a large score suggesting less peripheral neuropathy symptoms
Time Frame: Up to 52 weeks
Population: Patients that provided baseline and ≥ 1 follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Letrozole, Tamoxifen, Paclitaxel, PLD, Topotecan) | Arm B (Trametinib)
Number analyzed (Participants) | 98 | 100
score on a scale
  Baseline | 13.2 (3.5) | 12.8 (3.8)
  12 Weeks | 12.5 (4.0) | 12.6 (4.2)
  24 Weeks | 12.4 (4.0) | 12.1 (4.2)
  36 Weeks | 12.3 (3.8) | 12.6 (3.9)
  52 Weeks | 12.8 (3.2) | 12.4 (4.2)

7. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the number of months between study enrollment and documentation of disease progression (RECIST 1.1) or death from any cause. Patients still alive and disease free at the last followup were censored on the date of last CT Scan. RECIST v1.1 defines progression as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Time from study entry to time of progression or death, an average of 7 months for SOC and 13 months for the treatment (Trametinib) arm.
Population: Patients with sufficient tissue for analysis
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (Trametinib): KRAS/BRAF/NRAS mutant group (MAPK pathway) (Trametinib treatment) - Whole Exome Sequencing
- KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (SOC): KRAS/BRAF/NRAS mutant group (MAPK pathway) (Standard of Care treatment) - Whole Exome Sequencing
- KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (Trametinib): KRAS/BRAF/NRAS wild-type (MAPK pathway) (Trametinib treatment) - Whole Exome Sequencing
- KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (SOC): KRAS/BRAF/NRAS wild-type (MAPK pathway) (Standard of Care treatment) - Whole Exome Sequencing
Arm/Group | KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (Trametinib) | KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (SOC) | KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (Trametinib) | KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (SOC)
Number analyzed (Participants) | 22 | 22 | 48 | 42
Months | 13.2 [9.4 to 20.8] | 11.4 [3.7 to 13.3] | 7.3 [5.6 to 12.7] | 6.3 [3.7 to 9.9]
Statistical Analysis 1: Comparison: KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (Trametinib) vs KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (SOC); Test type: Superiority; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.28 to 1.07] — Estimation of treatment effect; Trametinib vs. SOC among patients with a mutation
Statistical Analysis 2: Comparison: KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (Trametinib) vs KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (SOC); Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.39 to 1.03] — Estimation of treatment effect; Trametinib vs. SOC among wild-type patients
Statistical Analysis 3: Comparison: KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (SOC) vs KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (SOC); Prognostic effect of the mutation status among patients in the SOC arm; Test type: Superiority; p = 0.0929, Chi-squared; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.34 to 1.08] — Estimation of mutation effect; mutant vs. wild-type in the SOC group
Statistical Analysis 4: Comparison: KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (Trametinib) vs KRAS/BRAF/NRAS Mutant Group (MAPK Pathway) (SOC) vs KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (Trametinib) vs KRAS/BRAF/NRAS Wild-type (MAPK Pathway) (SOC); Predictive effect biomarker p-value; Test type: Superiority; p = 0.7195, Chi-squared

8. Secondary Outcome: pERK Expression
Description: Will be quantified using the H-score derived from the immunohistochemistry analysis of patient tumor tissue and is expected to present as a continuous measure. will consider the prognostic and predictive abilities of pERK relative to objective response rate (ORR) or PFS. Analysis of the dichotomous markers will be supported by Kaplan Meier plots, and forest plots of the odds-ratio and hazard ratio estimates. Duration of response will be depicted using swimmer plots, with median duration estimated using Kaplan Meier methods. The multivariable models will include covariate adjustment for geographic region, performance status and number of prior regimens, presented using effect coding. The adjusted hazard- and odds- ratio estimates from the multivariable models will be supported by nominal p-values and 2-sided, 95% confidence intervals. Confidence intervals will be interpreted as the plausible range of values for the true (unobserved) ratio that is supported by the data.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Starting with the first treatment received, and ending 100 days after the last treatment, or at the last following, whichever is sooner. Time frame was approximately 30 months.
Groups:
- Crossover From Control to Experimental Arm: Patients randomized to the control arm who crossed over to the experimental arm after disease progression.
Arm/Group | Arm A - Control Arm | Arm B - Experimental Arm | Crossover From Control to Experimental Arm
All-Cause Mortality (participants affected / at risk) | 60/127 | 51/127 | 3/88
Serious Adverse Events (participants affected / at risk) | 43/127 | 45/127 | 25/88
Other Adverse Events (participants affected / at risk) | 124/127 | 127/127 | 88/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Control Arm (N=127) | Arm B - Experimental Arm (N=127) | Crossover From Control to Experimental Arm (N=88)
Anemia (Blood and lymphatic system disorders) | 1 | 4 | 1
Eye Disorders - Other (Eye disorders) | 2 | 2 | 0
Retinal Vascular Disorder (Eye disorders) | 0 | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 4 | 0 | 5
Colonic Stenosis (Gastrointestinal disorders) | 0 | 1 | 1
Colonic Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 11 | 3
Abdominal Pain (Gastrointestinal disorders) | 10 | 2 | 2
Mucositis Oral (Gastrointestinal disorders) | 1 | 1 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Jejunal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 1
Flu Like Symptoms (General disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Edema Limbs (General disorders) | 1 | 0 | 0
Death Nos (General disorders) | 1 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Infections And Infestations - Other (Infections and infestations) | 1 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1
Lung Infection (Infections and infestations) | 1 | 2 | 0
Kidney Infection (Infections and infestations) | 2 | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 6 | 2
Intestinal Stoma Obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ejection Fraction Decreased (Investigations) | 1 | 2 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0
Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 0 | 1 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 3 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 4 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Control Arm (N=127) | Arm B - Experimental Arm (N=127) | Crossover From Control to Experimental Arm (N=88)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 1 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 54 | 66 | 51
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Conduction Disorder (Cardiac disorders) | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 4 | 1
Palpitations (Cardiac disorders) | 5 | 5 | 0
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 2 | 0
Acute Coronary Syndrome (Cardiac disorders) | 2 | 0 | 1
Pulmonary Valve Disease (Cardiac disorders) | 0 | 1 | 0
Tricuspid Valve Disease (Cardiac disorders) | 0 | 2 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1 | 1
Cardiac Disorders - Other (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 8 | 7
Mitral Valve Disease (Cardiac disorders) | 0 | 1 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 4 | 1
Hearing Impaired (Ear and labyrinth disorders) | 2 | 2 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 3 | 2
Hypothyroidism (Endocrine disorders) | 2 | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0
Eye Disorders - Other (Eye disorders) | 0 | 1 | 0
Watering Eyes (Eye disorders) | 2 | 3 | 2
Keratitis (Eye disorders) | 1 | 1 | 0
Eye Pain (Eye disorders) | 3 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 2
Photophobia (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 3 | 2
Retinal Tear (Eye disorders) | 0 | 1 | 0
Retinopathy (Eye disorders) | 1 | 0 | 1
Corneal Ulcer (Eye disorders) | 0 | 1 | 0
Retinal Vascular Disorder (Eye disorders) | 0 | 2 | 0
Blurred Vision (Eye disorders) | 12 | 32 | 13
Dry Eye (Eye disorders) | 7 | 13 | 11
Retinal Detachment (Eye disorders) | 0 | 2 | 2
Floaters (Eye disorders) | 0 | 4 | 4
Eyelid Function Disorder (Eye disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 8 | 13 | 5
Dry Mouth (Gastrointestinal disorders) | 5 | 19 | 22
Colonic Obstruction (Gastrointestinal disorders) | 6 | 1 | 7
Colonic Stenosis (Gastrointestinal disorders) | 1 | 1 | 2
Colonic Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 2
Colonic Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 49 | 54 | 31
Diarrhea (Gastrointestinal disorders) | 43 | 92 | 53
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 44 | 58 | 33
Bloating (Gastrointestinal disorders) | 21 | 21 | 18
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Stomach Pain (Gastrointestinal disorders) | 1 | 3 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 9 | 15 | 9
Abdominal Pain (Gastrointestinal disorders) | 60 | 56 | 48
Rectal Hemorrhage (Gastrointestinal disorders) | 4 | 3 | 6
Oral Dysesthesia (Gastrointestinal disorders) | 0 | 2 | 4
Mucositis Oral (Gastrointestinal disorders) | 23 | 46 | 24
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Ileus (Gastrointestinal disorders) | 1 | 0 | 2
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 2 | 1
Oral Pain (Gastrointestinal disorders) | 1 | 5 | 4
Abdominal Distension (Gastrointestinal disorders) | 6 | 6 | 5
Nausea (Gastrointestinal disorders) | 65 | 77 | 48
Gastroparesis (Gastrointestinal disorders) | 0 | 1 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 10 | 11 | 10
Rectal Pain (Gastrointestinal disorders) | 0 | 2 | 0
Gastric Fistula (Gastrointestinal disorders) | 0 | 1 | 0
Fecal Incontinence (Gastrointestinal disorders) | 3 | 1 | 2
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 4 | 3
Ascites (Gastrointestinal disorders) | 7 | 5 | 2
Toothache (Gastrointestinal disorders) | 2 | 1 | 1
Jejunal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 3 | 1
Flatulence (Gastrointestinal disorders) | 2 | 4 | 4
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Pain (General disorders) | 13 | 25 | 13
Neck Edema (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 4 | 3
Localized Edema (General disorders) | 0 | 6 | 7
Irritability (General disorders) | 1 | 1 | 0
Flu Like Symptoms (General disorders) | 4 | 5 | 1
Edema Trunk (General disorders) | 1 | 3 | 1
Non-Cardiac Chest Pain (General disorders) | 6 | 7 | 3
Edema Limbs (General disorders) | 15 | 61 | 36
Edema Face (General disorders) | 1 | 10 | 5
Fatigue (General disorders) | 75 | 92 | 59
Fever (General disorders) | 13 | 22 | 12
Chills (General disorders) | 3 | 15 | 10
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Allergic Reaction (Immune system disorders) | 1 | 8 | 0
Infections And Infestations - Other (Infections and infestations) | 1 | 1 | 0
Wound Infection (Infections and infestations) | 4 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 6 | 14 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0
Vulval Infection (Infections and infestations) | 1 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 2 | 1 | 2
Skin Infection (Infections and infestations) | 6 | 19 | 10
Sinusitis (Infections and infestations) | 3 | 7 | 1
Sepsis (Infections and infestations) | 1 | 4 | 3
Rhinitis Infective (Infections and infestations) | 0 | 1 | 1
Rash Pustular (Infections and infestations) | 1 | 4 | 4
Pharyngitis (Infections and infestations) | 2 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1 | 0
Papulopustular Rash (Infections and infestations) | 0 | 12 | 1
Nail Infection (Infections and infestations) | 1 | 4 | 0
Mucosal Infection (Infections and infestations) | 1 | 2 | 1
Lung Infection (Infections and infestations) | 2 | 3 | 9
Laryngitis (Infections and infestations) | 0 | 4 | 0
Kidney Infection (Infections and infestations) | 2 | 3 | 1
Paronychia (Infections and infestations) | 0 | 11 | 9
Eye Infection (Infections and infestations) | 1 | 4 | 1
Device Related Infection (Infections and infestations) | 0 | 1 | 0
Small Intestine Infection (Infections and infestations) | 0 | 1 | 0
Gum Infection (Infections and infestations) | 1 | 0 | 0
Vaginal Infection (Infections and infestations) | 2 | 8 | 2
Urinary Tract Infection (Infections and infestations) | 18 | 29 | 14
Bronchial Infection (Infections and infestations) | 1 | 2 | 1
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 1
Lip Infection (Infections and infestations) | 0 | 1 | 0
Anorectal Infection (Infections and infestations) | 0 | 2 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urostomy Obstruction (Injury, poisoning and procedural complications) | 1 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intestinal Stoma Site Bleeding (Injury, poisoning and procedural complications) | 1 | 1 | 1
Intestinal Stoma Obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 2
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 7 | 0
Intestinal Stoma Leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 6 | 0
Weight Loss (Investigations) | 5 | 8 | 9
Weight Gain (Investigations) | 2 | 8 | 2
Platelet Count Decreased (Investigations) | 13 | 22 | 8
Lymphocyte Count Increased (Investigations) | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 6 | 4 | 2
Lipase Increased (Investigations) | 0 | 1 | 0
Inr Increased (Investigations) | 1 | 1 | 1
Ggt Increased (Investigations) | 1 | 1 | 2
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 2 | 2
Ejection Fraction Decreased (Investigations) | 1 | 10 | 7
Creatinine Increased (Investigations) | 10 | 25 | 15
Cholesterol High (Investigations) | 0 | 2 | 0
Neutrophil Count Decreased (Investigations) | 19 | 21 | 12
Cardiac Troponin I Increased (Investigations) | 0 | 2 | 0
Cpk Increased (Investigations) | 0 | 2 | 0
Cd4 Lymphocytes Decreased (Investigations) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 2 | 0
White Blood Cell Decreased (Investigations) | 21 | 28 | 17
Aspartate Aminotransferase Increased (Investigations) | 15 | 47 | 27
Alkaline Phosphatase Increased (Investigations) | 11 | 31 | 15
Alanine Aminotransferase Increased (Investigations) | 13 | 27 | 15
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 4 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 9 | 4
Hyponatremia (Metabolism and nutrition disorders) | 11 | 16 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 29 | 41 | 28
Hypokalemia (Metabolism and nutrition disorders) | 16 | 27 | 11
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 5 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 25 | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 | 42 | 24
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 8 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 5 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 25 | 32 | 16
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 10 | 11 | 7
Anorexia (Metabolism and nutrition disorders) | 24 | 33 | 35
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9 | 9 | 6
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 16 | 10
Muscle Weakness Trunk (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 10 | 6
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 24 | 24 | 20
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 11 | 15
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 4 | 1
Stroke (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 28 | 36 | 17
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 5 | 0
Paresthesia (Nervous system disorders) | 6 | 3 | 5
Memory Impairment (Nervous system disorders) | 6 | 6 | 4
Lethargy (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 24 | 28 | 20
Dysphasia (Nervous system disorders) | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 11 | 8
Sinus Pain (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 3 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 7 | 22 | 11
Concentration Impairment (Nervous system disorders) | 1 | 1 | 2
Cognitive Disturbance (Nervous system disorders) | 1 | 2 | 1
Personality Change (Psychiatric disorders) | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 24 | 16 | 17
Depression (Psychiatric disorders) | 11 | 26 | 10
Confusion (Psychiatric disorders) | 1 | 3 | 3
Anxiety (Psychiatric disorders) | 12 | 15 | 11
Agitation (Psychiatric disorders) | 1 | 3 | 0
Urine Discoloration (Renal and urinary disorders) | 1 | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 2 | 8 | 4
Urinary Tract Obstruction (Renal and urinary disorders) | 2 | 5 | 3
Urinary Retention (Renal and urinary disorders) | 2 | 4 | 5
Urinary Incontinence (Renal and urinary disorders) | 5 | 10 | 5
Urinary Tract Pain (Renal and urinary disorders) | 6 | 10 | 2
Urinary Frequency (Renal and urinary disorders) | 9 | 10 | 9
Proteinuria (Renal and urinary disorders) | 2 | 7 | 3
Hematuria (Renal and urinary disorders) | 3 | 20 | 4
Cystitis Noninfective (Renal and urinary disorders) | 2 | 1 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 3 | 1 | 2
Bladder Spasm (Renal and urinary disorders) | 1 | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 0 | 4
Vaginal Pain (Reproductive system and breast disorders) | 1 | 2 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 8 | 3 | 6
Vaginal Fistula (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 4 | 5 | 2
Uterine Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 5 | 5 | 2
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 8 | 3 | 6
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 3 | 2 | 2
Breast Pain (Reproductive system and breast disorders) | 2 | 0 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 8
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 6
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 15 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 | 44 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 30 | 19
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 6 | 2
Skin Ulceration (Skin and subcutaneous tissue disorders) | 2 | 8 | 5
Skin Induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 3 | 4
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 13 | 80 | 50
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 25 | 18
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Periorbital Edema (Skin and subcutaneous tissue disorders) | 0 | 6 | 4
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 21 | 8 | 10
Pain Of Skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 28 | 54 | 30
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 1 | 2 | 4
Nail Discoloration (Skin and subcutaneous tissue disorders) | 3 | 4 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 4 | 3
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 17 | 56 | 40
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 28 | 21
Thromboembolic Event (Vascular disorders) | 6 | 11 | 4
Lymphedema (Vascular disorders) | 3 | 5 | 1
Hypotension (Vascular disorders) | 2 | 5 | 3
Hypertension (Vascular disorders) | 27 | 49 | 30
Hot Flashes (Vascular disorders) | 35 | 14 | 13
Flushing (Vascular disorders) | 3 | 3 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Genital Edema (Reproductive system and breast disorders) | 0 | 0 | 1
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 2
Heart Failure (Cardiac disorders) | 0 | 0 | 1
Flashing lights (Eye disorders) | 0 | 0 | 1
Chest pain - Cardiac (Cardiac disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 1
Esophageal Stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Multi-Organ failure (General disorders) | 0 | 0 | 1
Bladder infection (Infections and infestations) | 0 | 0 | 1
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
The pERK expression analysis is still under development, and will not be available for approximately 2 - 3 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT02101788/Prot_SAP_001.pdf